CLINICAL TRIAL: NCT00653159
Title: Intrauterine Contraception for Adolescents Aged 14 to 18: A Multi-center Randomized Controlled Feasibility Trial of Levonorgestrel-releasing Intrauterine System Compared to the Copper T 380A
Brief Title: Maintaining Intrauterine Devices (IUDs) in Teens (MINT): A Randomization Trial
Acronym: MINT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15498A
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Contraception
Keywords: Intrauterine device, contraception, unplanned pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirena IUD [LNG-IUS] (Active Comparator): Participants in this arm had a Levonorgestrel-releasing intrauterine device (LNG-IUS), also known as the Mirena IUD, inserted within the first 5 days of the adolescent's menstrual cycle, at least 7 weeks after a vaginal or cesarean delivery or second-trimester abortion or at least 3 weeks after a first-trimester abortion. For participants who had used depot-medroxyprogesterone acetate, insertions occurred at least 6 months after the participant's last injection. Participants were blinded to the device type; however, investigators and research assistants were not.
  Interventions: Device: Levonorgestrel-releasing intrauterine device (LNG-IUS)
- Paragard IUD [Copper T380A] (Active Comparator): Participants in this arm had a Copper T380A intrauterine device (CuT380A), also known as the Paragard IUD, inserted within the first 5 days of the adolescent's menstrual cycle, at least 7 weeks after a vaginal or cesarean delivery or second-trimester abortion or at least 3 weeks after a first-trimester abortion. For participants who had used depot-medroxyprogesterone acetate, insertions occurred at least 6 months after the participant's last injection. Participants were blinded to the device type; however, investigators and research assistants were not.
  Interventions: Device: Copper T380A intrauterine device (CuT380A)

INTERVENTIONS:
Device: Levonorgestrel-releasing intrauterine device (LNG-IUS) — Teens are randomly assigned to receive the LNG-IUS after completing a screening visit.
  Other Names: Mirena IUD
  Arms: Mirena IUD [LNG-IUS]
Device: Copper T380A intrauterine device (CuT380A) — Teens are randomly assigned to Copper T380 after the screening visit
  Other Names: Paraguard IUD
  Arms: Paragard IUD [Copper T380A]

SUMMARY:
This is a pilot study to determine the feasibility for a randomized controlled trial of two forms of intrauterine contraception: the Levonorgestrel intrauterine system (LNG-IUS) and the Copper T 380A.

DETAILED DESCRIPTION:
Teenagers have the highest percentage of unintended pregnancies, and often struggle to comply with daily methods of contraception. The intrauterine device (IUD) provides safe, long-term protection and rates highly for patient satisfaction. It also does not require repeat prescriptions or clinic visits, making it a potentially attractive method among teens. However, in adolescent populations, there is both a lack of information about the IUD, as well as few studies that have examined the use of these devices. This study will examine whether a larger scale study on this topic is feasible. IT will address the feasibility of recruiting, consenting, screening, enrolling, randomizing, and retaining adolescents randomized to the LNG-IUS or Copper T 380a.

ELIGIBILITY:
Inclusion Criteria:

Healthy, sexually active females age 14 to 18 who:

* Are interested in long term, reversible contraception
* Have regular menstrual cycles (21-35 days)
* Are not planning a pregnancy within the next 6 months

Exclusion Criteria:

Sexually active females age over the age of 18 or who:

* Are not interested in long term, reversible contraception
* Do not have regular menstrual cycles (21-35 days)
* Are planning a pregnancy within the next 6 months

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, Principal Investigator — The University of Chicago Medicine
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted within the Section of Family Planning in the Department of Obstetrics and Gynecology at The University of Chicago and within the Department of Family Medicine at the University of Illinois-Chicago. From December 2007 through June 2008, 37 adolescent females were approached regarding the study.
Pre-assignment Details: All of the 23 enrolled subjects were ultimately randomized to the treatment arms (12 to LNG-IUS and 11 to CuT380A).
Groups:
- Paragard IUD [CuT380A]: Paragard intrauterine device (IUD), Copper T 380A
- Mirena IUD [LNG-IUS]: Mirena intrauterine device (IUD), Levonorgestrel Intrauterine System
Period: Overall Study
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Started | 11 | 12
Completed | 6 | 9
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS] | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Median (Full Range); unit: years] | 17 [15 to 18] | 16.5 [14 to 18] | 16.5 [14 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 4 | 2 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Education [Number; unit: participants]
  8th grade or less | 0 | 1 | 1
  Current high school student | 8 | 10 | 18
  High school diploma/GED | 2 | 0 | 2
  Some college/current college student | 1 | 1 | 2
Parous [Number; unit: participants] — A parous female participant has given birth one or more times. A female is nulliparous if she has never given birth.
  participants
    Parous | 7 | 4 | 11
    Nulliparous | 4 | 8 | 12
Previous STI [Number; unit: participants] — Number of participants who have previously tested positive for one or more of the following sexually transmitted infections (STI) during the screening visit: chlamydia, gonorrhea, trichomonas, and vaginal warts.
  participants
    Yes | 4 | 2 | 6
    No | 7 | 10 | 17
Presence of STI at screening visit [Number; unit: participants] — Number of participants who tested positive for one or more of the following sexually transmitted infections (STI) during the screening visit: chlamydia, gonorrhea, trichomonas, and vaginal warts.
  participants
    Yes | 1 | 3 | 4
    No | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Percentage of participants who completed the final visit (i.e., not subject to early termination or loss to follow-up)
Time Frame: 6 months
Population: All study participants were included in the analysis.
Measure: Number; unit: percentage of randomized subjects
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Number analyzed (Participants) | 11 | 12
percentage of randomized subjects | 55 | 75
Statistical Analysis 1: Comparison: Paragard IUD [CuT380A] vs Mirena IUD [LNG-IUS]; Fisher's exact test was used to examine the significance of the association between IUD type (Paragard or Mirena) and whether or not the subject completed the final study visit at 6 months. Under the null hypothesis, study completion rates are similar for both IUD types; Test type: Superiority or Other; p = 0.4003, Fisher Exact; Two-sided test

2. Secondary Outcome: Heavy Bleeding Rates
Description: Rates of participants experiencing heavy bleeding among teens randomized to the LNG-IUS or Copper T 380A.
Time Frame: 6 months
Population: All study participants were included in the analysis.
Measure: Number; unit: percentage of randomized subjects
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Number analyzed (Participants) | 11 | 12
percentage of randomized subjects | 55 | 33
Statistical Analysis 1: Comparison: Paragard IUD [CuT380A] vs Mirena IUD [LNG-IUS]; Fisher's exact test was used to examine the significance of the association between IUD type (Paragard or Mirena) and whether or not the subject experienced heavy bleeding. Under the null hypothesis, heavy bleeding rates are similar for both IUD types; Test type: Superiority or Other; p = 0.4136, Fisher Exact; Two-sided test

3. Secondary Outcome: Pregnancy Rates
Description: Proportion of subjects who became pregnant within 6 months of IUD insertion
Time Frame: 6 months
Population: All study participants were included in the analysis.
Measure: Number; unit: percentage of randomized subjects
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Number analyzed (Participants) | 11 | 12
percentage of randomized subjects | 9 | 0
Statistical Analysis 1: Comparison: Paragard IUD [CuT380A] vs Mirena IUD [LNG-IUS]; Fisher's exact test was used to examine the significance of the association between IUD type (Paragard or Mirena) and whether or not the subject became pregnant within 6 months of IUD insertion. Under the null hypothesis, pregnancy rates are similar for both IUD types; Test type: Superiority or Other; p = 0.4783, Fisher Exact; Two-sided test

4. Secondary Outcome: Expulsion Rates
Description: Rates of partial or complete expulsion for teens randomized to the LNG-IUS or Copper T 380A. Patients experiencing partial expulsion had IUDs visible on speculum exam. Complete expulsion is characterized by complete evacuation of the IUD.
Time Frame: 6 months
Population: All study participants were included in the analysis.
Measure: Number; unit: percentage of randomized subjects
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Number analyzed (Participants) | 11 | 12
percentage of randomized subjects | 18 | 0
Statistical Analysis 1: Comparison: Paragard IUD [CuT380A] vs Mirena IUD [LNG-IUS]; Fisher's exact test was used to examine the significance of the association between IUD type (Paragard or Mirena) and whether or not the subject experienced expulsion of the IUD. Under the null hypothesis, expulsion rates are similar for both IUD types; Test type: Superiority or Other; p = 0.2174, Fisher Exact; Two-sided test

5. Secondary Outcome: Device Satisfaction Rates
Description: Satisfaction rate is the proportion of subjects who report being "happy" or "very happy" with their assigned intrauterine contraceptive method on the date of their 6 month study visit.
Time Frame: 6 months
Population: Only subjects who were not lost to follow-up at 6 months were included in this analysis.
Measure: Number; unit: percentage of subjects completing study
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Number analyzed (Participants) | 10 | 10
percentage of subjects completing study | 80 | 70
Statistical Analysis 1: Comparison: Paragard IUD [CuT380A] vs Mirena IUD [LNG-IUS]; Fisher's exact test was used to examine the significance of the association between IUD type (Paragard or Mirena) and whether or not the subject reported being satisfied ("happy" or "very happy") at the 6 month study visit. Under the null hypothesis, satisfaction rates are similar for both IUD types; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Two-sided test

ADVERSE EVENTS:
Arm/Group | Paragard IUD [CuT380A] | Mirena IUD [LNG-IUS]
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 11/11 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paragard IUD [CuT380A] (N=11) | Mirena IUD [LNG-IUS] (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 1 — Disorder characterized by reduction in the amt of hemoglobin in 100 ml of blood. Signs/symptoms may include pallor of the skin and mucous membranes, shortness of breath, palpitations of the heart, soft systolic murmurs, lethargy, and fatigability.
Abdominal pain (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by a sensation of marked discomfort in the abdominal region.
Bloating (Gastrointestinal disorders) | 2 | 2 — A disorder characterized by subject-reported feeling of uncomfortable fullness of the abdomen.
Vomiting (Gastrointestinal disorders) | 0 | 1 — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Nausea (Gastrointestinal disorders) | 0 | 1 — A disorder characterized by a queasy sensation and/or the urge to vomit.
Fatigue (General disorders) | 0 | 1 — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Fever (General disorders) | 2 | 3 — A disorder characterized by elevation of the body's temperature above the upper limit of normal.
Leg pain (General disorders) | 0 | 1 — Pain in the leg.
Abscess/infection of Bartholin's gland (Infections and infestations) | 0 | 1 — Abscess/infection of Bartholin's gland
Bacterial vaginosis (Infections and infestations) | 1 | 0 — Bacterial vaginosis is the name of a condition in women where the normal balance of bacteria in the vagina is disrupted and replaced by an overgrowth of certain bacteria. It is sometimes accompanied by discharge, odor, pain, itching, or burning.
Trichomoniasis (Infections and infestations) | 0 | 1 — Trichomoniasis (or "trich") is a very common sexually transmitted disease (STD) that is caused by infection with a protozoan parasite called Trichomonas vaginalis.
Urinary tract infection (Infections and infestations) | 1 | 0 — A disorder characterized by an infectious process involving the urinary tract, most commonly the bladder and the urethra
Weight gain (Investigations) | 1 | 2 — A finding characterized by an increase in overall body weight; for pediatrics, greater than the baseline growth curve.
Headaches (Nervous system disorders) | 1 | 1 — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve
Libido decreased (Psychiatric disorders) | 1 | 0 — A disorder characterized by a decrease in sexual desire.
Psychiatric disorders - Other (Mood Swings) (Psychiatric disorders) | 1 | 2 — A mood swing is an extreme or rapid change in mood.
Breast swelling (Reproductive system and breast disorders) | 1 | 2 — Swelling and tenderness of the breasts
Irregular menstruation (Reproductive system and breast disorders) | 1 | 1 — A disorder characterized by irregular cycle or duration of menses
Menorrhagia (Reproductive system and breast disorders) | 5 | 5 — A disorder characterized by abnormally heavy vaginal bleeding during menses.
Menstrual pain (Reproductive system and breast disorders) | 11 | 5 — Pain during menses
Vaginal discharge (Reproductive system and breast disorders) | 0 | 3 — A disorder characterized by vaginal secretions. Mucus produced by the cervical glands is discharged from the vagina naturally, especially during the childbearing years.
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 — A disorder characterized by inflammation involving the vagina. Symptoms may include redness, edema, marked discomfort and an increase in vaginal discharge
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 — Acne is a common human skin disease, characterized by areas of skin with seborrhea (scaly red skin), comedones (blackheads and whiteheads), papules (pinheads), pustules (pimples), nodules (large papules) and possibly scarring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes